CLINICAL TRIAL: NCT00914992
Title: Regulation of Optic Nerve Head Blood Flow During Combined Changes in Intraocular Pressure and Arterial Blood Pressure.
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Sponsor: Medical University of Vienna (Other)
Responsible Party: Elzbieta Polska, MD, Department of Clinical Pharmacology, Medical University of Vienna
Allocation: Non-Randomized | Model: Crossover | Masking: None | Purpose: Basic Science
Other Study IDs: OPHT-310505
Record Dates: First submitted 2009-06-03; First posted 2009-06-05 (Estimated); Last update posted 2014-12-08 (Estimated); Status verified 2014-11

CONDITIONS: Healthy
Keywords: optic disk; regional blood flow; autoregulation

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

INTERVENTIONS:
Procedure: Suction cup application — The IOP will be raised by an 11 mm diameter, standardized suction cup placed on the temporal sclera with the anterior edge at least 1 mm from the limbus.
Other: Squatting — Squatting

SUMMARY:
Autoregulation is the ability of a vascular bed to maintain blood flow despite changes in perfusion pressure. The existence of an effective autoregulation in the optic nerve head (ONH) circulation has been shown in animals and humans. Moderate elevation of intraocular pressure (IOP) caused only slight effect on ONH blood flow in monkeys, cats and rabbits. In humans, during an artificial IOP rise using a suction cup method the ONH blood flow maintains almost constant until IOP reaches 40-55 mmHg. During isometric exercise the upper limit of autoregulation appears to be approximately 40% above the baseline ocular perfusion pressure. The mechanism behind ONH blood flow autoregulation is still unknown. The present experiments are designed to improve the investigators' knowledge of the physiology of regulatory mechanisms in ONH circulation, which may be helpful for a better understanding of blood flow abnormalities in glaucoma. This is of importance, because there is increasing evidence that vascular dysregulation plays a role in the development of glaucomatous damage.

ELIGIBILITY:
Inclusion Criteria:

* Men aged between 19 and 35 years, nonsmokers
* Body mass index between 15th and 85th percentile
* Normal findings in the medical history and physical examination unless the investigator considers an abnormality to be clinically irrelevant
* Normal ophthalmic findings, ametropia < 1 Dpt

Exclusion Criteria:

* Regular use of medication, abuse of alcoholic beverages, participation in a clinical trial in the 3 weeks preceding the study
* Treatment in the previous 3 weeks with any drug
* Symptoms of a clinically relevant illness in the 3 weeks before the first study day
* Blood donation during the previous 3 weeks
* Presence of intraocular pathology: ocular hypertension, glaucoma, retinal vasculopathy or other retinal diseases

Ages: 19 Years to 35 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 0 (Actual)
Dates: Start 2009-07; Primary Completion 2010-12 (Actual); Study Completion 2010-12 (Actual)

PRIMARY OUTCOMES:
Ocular perfusion pressure - ONH blood flow relationship | 9 months

CONTACTS AND LOCATIONS:
Overall Officials: Elzbieta Polska, MD, Study Director — Department of Clinical Pharmacology, Medical University of Vienna
Locations (1):
- Department of Clinical Pharmacology, Medical University of Vienna, Vienna, Austria